CLINICAL TRIAL: NCT03014544
Title: A Randomized, Multicenter, Crossover Study to Assess the Performance Validity and Test-Retest Reliability of a Computer-Administered Cognitive Test Battery in Subjects With Major Depressive Disorder
Brief Title: Study to Evaluate the Performance Validity and Test-Retest Reliability of a Computer-Administered Cognitive Test Battery in Participants With Major Depressive Disorder (MDD)
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108211; NOPRODMDD0003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-11-18; First posted 2017-01-09 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Group 1: Sequence AABB: Participants of main study with Major Depressive Disorder (MDD) will be assigned in test sequence group AABB (Group 1) to undergo sequential cognitive performance evaluations by Test A (Computer- administered test battery) on Test Day 1 (Study Day 1) and Test Day 2 (Study Day 15 to 22) followed by Test B (Examiner-administered test battery) on Test Day 3 (Study Day 29 to 43) and Test Day 4 (Study Day 43 to 64). Each separated by a memory washout period of 14 to 21 days.
  Interventions: Device: Computer- administered test battery; Device: Examiner- administered test battery
- Group 2: Sequence BBAA: Participants of main study with MDD will be assigned in test sequence group BBAA (Group 2) to undergo sequential cognitive performance evaluations by Test B (Examiner-administered test battery) on Test Day 1 (Study Day 1) and Test Day 2 (Study Day 15 to 22) followed by Test A (Computer- administered test battery) on Test Day 3 (Study Day 29 to 43) and Test Day 4(Study Day 43 to 64). Each separated by a memory washout period of 14 to 21 days.
  Interventions: Device: Computer- administered test battery; Device: Examiner- administered test battery

INTERVENTIONS:
Device: Computer- administered test battery — Participants in this observational study will only undergo sequential cognitive performance evaluations by computer- administered cognitive test battery.
  Other Names: REVERE.D
Device: Examiner- administered test battery — Participants in this observational study will only undergo sequential cognitive performance evaluations by examiner- administered cognitive test battery.

SUMMARY:
The purpose of this study is to examine concurrent validity of 8 computerized tests intended for the assessment of cognitive function in participants with Major Depressive Disorder (MDD), relative to 8 corresponding and previously validated examiner-administered cognitive tests.

ELIGIBILITY:
Inclusion Criteria:

* a) Substudy A and Main Study:
* Primary diagnosis of Major depressive disorder (MDD), made or confirmed by the investigator according to the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) criteria
* Demonstrated an adequate clinical response within the past 24 months, and is currently maintaining this response, to a stable oral antidepressant treatment regimen of no more than 2 of the following: selective serotonin reuptake inhibitor (SSRI), serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressants, in any formulation (fluvoxamine, citalopram, duloxetine, escitalopram, fluoxetine, milnacipran, levomilnacipran, paroxetine, sertraline, venlafaxine, desvenlafaxine, vilazodone, or vortioxetine), or bupropion antidepressants, without any dosing changes for the most recent 6 weeks. The dose and duration of treatment will be documented by the investigator using the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH-ATRQ) and verified against the available medical and pharmacy records or medication bottles/package labels
* Required to have a Montgomery-Asberg Depression Rating Scale (MADRS) total score of less than or equal (<=)17 at screening and baseline (Test Day 1) visits as well as less than or equal (<=)19 during subsequent testing days (main study). Participants are also required to have a Clinical Global Impression - Severity (CGI-S) total score of <=3 during testing days (main study)
* Must have adequate visual and hearing acuity to perform all aspects of the cognitive and functional assessments as determined during physical examination
* b) Substudy B (Healthy Participants):
* Must be healthy on the basis of physical examination, vital signs examination, and medical history performed at screening. This determination must be recorded in the participant's source documents and initialed by the investigator
* Body mass index (weight [kilogram (kg)]/height^2 [meter (m)]^2) between 18 and 30 kg/m2 (inclusive)
* Blood pressure (after the participant is sitting for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) inclusive, systolic, and no higher than 90 mmHg diastolic
* Must sign an Informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

* a) Substudy A and Main Study:
* Has any of the following acute or chronic psychiatric conditions, according to Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) criteria: Major depressive disorder (MDD) with psychotic features (lifetime), bipolar disorder (including lifetime diagnosis), obsessive-compulsive disorder, post-traumatic stress disorder, borderline personality disorder, anorexia nervosa, schizophrenia, schizoaffective disorder, or minor and major neurocognitive disorders (including dementia)
* History of any acute or chronic neurological condition (for example (eg), stroke, epilepsy, Parkinson's disease)
* b) Substudy B (Healthy Participants):
* History of drug or alcohol abuse, with a severity of at least moderate or severe, according to DSM-5 criteria, within 6 months before screening or positive test result(s) for alcohol or drugs of abuse (including barbiturates, opiates, cocaine, cannabinoids, amphetamines and benzodiazepines) at screening or admission on Day 1
* Participant has clinically significant liver or renal insufficiency; cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances. A significant primary sleep disorder is exclusionary, including primary insomnia and hypersomnia, narcolepsy, breathing-related sleep disorders, circadian-rhythm sleep disorders, and dyssomnias not otherwise specified
* Has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (for example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants enrolled in substudy A and main study will be man or woman with major depressive disorder (MDD) and participants enrolled in substudy B will be healthy participants to evaluate cognitive performance at the clinic site.
Sampling Method: Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Performance Score on a Cognitive Test Battery Evaluated by Symbol Sorting Test (SST) | Up to Test Day 4 (Day 43 to 64)
  The SST is designed as a measure of executive function. The SST requires the participant to sort symbols, based on symbol features such as color, shape, and number. No sorting criteria are provided to participants, rather the participant is provided feedback whether his/her response is correct or incorrect. Responses will be scored for Categories Achieved and Percent Perseverative Errors by computerized cognitive test battery.
Performance Score on a Cognitive Test Battery Evaluated by Digit Span Forward Test (DSFT) | Up to Test Day 4 (Day 43 to 64)
  The DSFT is a widely used measure of attention and working memory, with versions included in a number of cognitive test batteries. The DSFT measures aspects of attention (freedom from distractibility) and working memory, and has been shown to be impaired in participants with MDD. The participant is asked to repeat a sequence of digits in the order presented. Participant will respond by pressing the keys on a keypad that correspond to the digits recalled. Two points will be given if the participant moves to the next sequence of digits with 1 attempt; 1 point will be given if the participant moves to the next sequence with 2 attempts; and 0 points will be given if the participant fails both attempts for a particular span. The score is the sum of correct responses. The length of the longest span of digits recalled will be used as a secondary score (up to 9).
Performance Score on a Cognitive Test Battery Evaluated by Digit Span Backward Test (DSBT) | Up to Test Day 4 (Day 43 to 64)
  The DSBT is a widely used measure of attention and working memory, with versions included in a number of cognitive test batteries. The DSBT is thought to be a more complex span task than the DSFT as it also measures spatial/visual processing, and has been shown to be impaired in participants with MDD. The participant is asked to repeat a sequence of digits in reverse from the order presented. Participant will respond by pressing the keys on a keypad that correspond to the digits recalled in reverse order. Two points will be given if the participant moves to the next sequence of digits with 1 attempt; 1 point will be given if the participant moves to the next sequence with 2 attempts; and 0 points will be given if the participant fails both attempts for a particular span. The score is the sum of correct responses. The length of the longest span of digits recalled (backwards) will be used as a secondary score (up to 8).
Performance Score on a Cognitive Test Battery Evaluated by Word List Recall Test (WLRT) | Up to Test Day 4 (Day 43 to 64)
  The WLRT used for the computerized test battery that measures person's ability to encode, consolidate, store, and retrieve verbal information and is a sensitive test of verbal learning and memory in a variety of disease states, including MDD. The memory test will include a list of 15 words presented aloud, one at a time, through the iPad. After the 15-word list is presented, the participant will be asked to verbally recall as many of the words as possible. The 15 word list and participant recall will be conducted 4 more times (total 5 times). After the 5th learning trial and recall, performance on the learning trials of the original word list and on the delayed recall will be considered as the primary scores. The participant's responses during the WLRT will be recorded and scored using 2 methods: by the speech recognition engine (SRE) and by an on-site test supervisor who will record the responses directly on the Revere.D application from a touch screen on the iPad.
Performance Score on a Cognitive Test Battery Evaluated by Visuospatial Block Recall Test (VBRT) | Up to Test Day 4 (Day 43 to 64)
  The VBRT is based on a visuospatial learning test that requires participants to recall the location of colored tiles within an onscreen grid. Performance on visuospatial recall tasks has been shown to be lowered in anxious, depressed, or older healthy participants, as well as in participants with mild traumatic brain injury, schizophrenia, and acquired immune deficiency syndrome (AIDS) dementia complex. The participant is shown a sequence of on screen grids on which an increasingly complex pattern of colored tiles is depicted. Each pattern displays for only a brief period (0.5 seconds), after which participants are asked to recall the pattern. Recall accuracy (the number of correctly recalled patterns) is recorded by computerized cognitive test battery.
Performance Score on a Cognitive Test Battery Evaluated by Symbol Digit Matching Test (SDMaT) | Up to Test Day 4 (Day 43 to 64)
  The SDMaT measures the time to pair abstract symbols with specific numbers. The test includes a coding key consisting of 9 abstract symbols, each paired with a number ranging from 1 to 9. Following the key, the participant is presented with randomly ordered symbols and is required to enter the number corresponding to each symbol as fast as possible using a keypad. The number of correct digit entries within 90 seconds is recorded by computerized cognitive test battery .
Performance Score on a Cognitive Test Battery Evaluated by Trail Making Test Form B (TMT-B) | Up to Test Day 4 (Day 43 to 64)
  The computerized (Revere.D) version of the TMT-B is modeled after the paper-and-pencil version of the test. The TMT-B measures divided attention and executive function (tracking and sequencing). The participant is instructed to draw a line to connect a set of 25 consecutively numbered and lettered circles, alternating sequentially between numbers and letters (that is, 1 A 2 B). The participant is instructed to work as quickly as possible while still maintaining accuracy. The TMT-B has acceptable reliability; reliability coefficients have typically been reported as exceeding 0.65. The TMT-B is sensitive to cognitive decline associated with MDD.
Performance Score on a Cognitive Test Battery Evaluated by Block Maze Test (BMT) | Up to Test Day 4 (Day 43 to 64)
  The BMT used in this study is modeled after published maze learning tests, such as the Groton Maze Learning Test, that assess processing speed, working memory, spatial learning, and error monitoring. In the BMT, the participant learns over 13 trials to navigate a path across tiles from a starting position to a target position using a set of predefined rules. The primary measure is total number of errors made in the 3 trials; the total time required for correct completion of the 3 trials will be used as a secondary score that will be evaluated by computerized cognitive test battery.
Performance Score on a Cognitive Test Battery Evaluated by Rey Auditory Verbal Learning Test (RAVLT) | Up to Test Day 4 (Day 43 to 64)
  The RAVLT is a commonly used measure of a person's ability to encode, consolidate, store, and retrieve verbal information and is a sensitive test of verbal learning and memory in a variety of disease states, including MDD. The test will be administered by an examiner who will read the words aloud to the participant . The memory test will include a list of 15 words presented one at a time verbally by the examiner. After the 15-word list is presented, the participant will be asked to verbally recall as many of the words as possible. The 15 word list and participant recall will be conducted 4 more times (total 5 times). After the 5th learning trial and recall performance on the learning trials of the original word list and on the delayed recall will be considered as the primary scores that will be evaluated by examiner-administered cognitive test battery.
Performance Score on a Cognitive Test Battery Evaluated by Brief Visuospatial Memory Test-Revised (BVMT-R) | Up to Test Day 4 (Day 43 to 64)
  The BVMT-R is a test of visual learning and recall. Participants are presented with 6 geometric figures in a 2*3 visual array; presentation is on a sheet of paper for a 10 second exposure. Participants are asked to draw as many figures in their proper locations as they remember, for each of 3 learning trials. The test has good test-retest reliability; r [greater than (>)]0.96 for the learning trials. The BVMT-R is included in the MATRICS Consensus Cognitive Battery. The total recall score will be used in this study that will be evaluated by examiner-administered cognitive test battery.
Performance Score on a Cognitive Test Battery Evaluated by Symbol Digit Modalities Test (SDMT) | Up to Test Day 4 (Day 43 to 64)
  The SDMT is a widely used, paper-and-pencil assessment of complex scanning and visual tracking, requiring elements of attention, visuoperceptual processing, working memory, and cognitive/psychomotor speed.The test is viewed as a robust screening test for adult neuropsychological impairment and has been used to demonstrate worse cognitive functioning in patients with MDD. The SDMT measures the time to pair abstract symbols with specific numbers. The test includes a coding key consisting of 9 abstract symbols, each paired with a number ranging from 1 to 9. Following the key, the participant is presented with randomly ordered symbols and is required to write the number corresponding to each symbol as fast as possible. The number of correct substitutions within 90 seconds is recorded by examiner-administered cognitive test battery.
Performance Score on a Cognitive Test Battery Evaluated by Neuropsychological Assessment Battery - Maze Test (NAB-MT) | Up to Test Day 4 (Day 43 to 64)
  The NAB-MT is a test in which participants are asked to complete 7 increasingly complex paper-and-pencil mazes; scores include time to completion.The test assesses aspects of executive function, especially planning and foresight. It was standardized on a sample of more than 1,400 healthy adults. Extensive validation evidence has been established through exploratory and confirmatory factor analyses, criterion validity investigations, and several clinical validation studies. It has been used to demonstrate neurocognitive impairments in patients with depression. The NAB-MT is included in the MATRICS Consensus Cognitive Battery. The time to completion score will be used in this study that will be evaluated by examiner-administered cognitive test battery.
Performance Score on a Cognitive Test Battery Evaluated by Wisconsin Card Sorting Test (WCST) | Up to Test Day 4 (Day 43 to 64)
  WCST is a widely used measure of executive function. WCST requires the participant to sort symbols based on symbol features such as color, shape and number without providing instructions as to matching criteria; rather the participant is provided feedback whether a particular match is right or wrong. Responses will be scored for Categories Achieved and Percent Perseverative Errors by examiner-administered cognitive test battery.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (20):
- United States (20):
  - Birmingham, Alabama
  - Anaheim, California
  - Beverly Hills, California
  - Glendale, California
  - Long Beach, California
  - Temecula, California
  - Denver, Colorado
  - Hartford, Connecticut
  - Jacksonville, Florida
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Saint Charles, Missouri
  - Lincoln, Nebraska
  - Buffalo, New York
  - Mount Kisco, New York
  - New York, New York
  - Allentown, Pennsylvania
  - Dallas, Texas
  - Salt Lake City, Utah